CLINICAL TRIAL: NCT06677671
Title: Comparison of Exercise Capacity, Muscle Parameters and Quality of Life Parameters in Chronic Obstructive Pulmonary Disease Patients and Healthy Individuals
Brief Title: Comparison of Clinical Parameters in Chronic Obstructive Pulmonary Disease Patients and Healthy Individuals
Status: Active, not recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Cansu Özkılıçaslan, Physiotherapist, M.Sc, Hacettepe University
Other Study IDs: AEŞH-BADEK-2024-553
Record Dates: First submitted 2024-11-03; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: copd; exercise capacity; muscle parameters
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy: Healthy Individuals
- COPD: Chronic Obstructive Pulmonary Disease Patients

SUMMARY:
The investigators think that the functions of core stabilization muscles are different in chronic obstructive pulmonary disease (COPD) patients than in healthy individuals. This muscle group plays an important role not only in stabilization but also in respiratory parameters. No study has been found investigating the functions of these muscles in this patient group. The investigators aimed to compare respiratory parameters, muscle parameters, exercise capacity, balance, quality of life, anxiety and depression levels in individuals with COPD and healthy individuals.

DETAILED DESCRIPTION:
Individuals diagnosed with COPD between the ages of 40-80 who applied to Ankara Etlik City Hospital Chest Diseases Polyclinic will be included in the study. Healthy individuals will be between the ages of 40-80 who volunteered to participate in the study. Data collection tools will be made by the same researchers.

For calculating the sample size required for the study, a power analysis will be conducted using pilot data after evaluating 10 individuals with COPD and 10 healthy adults.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Individuals with COPD:

* Being diagnosed with COPD
* Being between the ages of 40-80
* Being clinically stable (not having had an exacerbation in the last month)
* Being able to cooperate with the tests
* Not participating in any exercise training studies
* Being willing to participate in the study

Inclusion Criteria for Healthy Individuals:

* Being between the ages of 40-80
* Not having a known acute or chronic health problem that would prevent the performance of the tests or affect the performance of the tests
* Not participating in any exercise training program
* Being willing to participate in the study

Exclusion Criteria:

Exclusion Criteria for Individuals with COPD:

* Having other lung or lung involvement diseases other than COPD
* Having uncontrolled hypertension, arrhythmia and a history of myocardial infarction in the last month, unstable angina, advanced heart failure and other cardiac instability conditions
* Being hemodynamically unstable
* Being on noninvasive mechanical ventilation (NIMV) and long-term oxygen therapy (LTOT)
* Having a history of neuromuscular disease, scoliosis, chest wall surgery
* Having pregnancy and malignancy
* Having orthopedic or surgical conditions that would prevent participation in tests
* Not willing to participate in the study

Exclusion Criteria for Healthy Individuals:

* Having a known acute or chronic health problem that would prevent the performance of the tests or affect the performance of the tests
* Being pregnant
* Not willing to participate in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients and volunteer healthy individuals admitted to Ankara Etlik City Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-07-18 (Estimated); Study Completion 2026-07-18 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise test | September 2024, July 2026
  Cardiopulmonary exercise test will be performed to evaluate the exercise capacity of the individuals who will participate in the study. During the test, individuals' respiratory and cardiac parameters will be recorded.

SECONDARY OUTCOMES:
Respiratory function | September 2024, July 2026
  Respiratory functions will be assessed using spirometry (Cosmed Microquark-PC Based Spirometer, Rome, Italy) according to the criteria of the European Respiratory Society (ERS) and the American Thoracic Society (ATS).
Respiratory muscle strength | September 2024, July 2026
  Respiratory muscle strength will be assessed with a portable, electronic oral pressure measuring device (Cosmed Pony Fx, Milan, Italy). Respiratory muscle strength will be determined by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP). Percentage of expected reference values according to gender and age will be used for the MIP value. The clinical significance for this patient group is 17.2 cmH2O for the measured MIP value.
Muscle activity and muscle thickness | September 2024, July 2026
  In our study, muscle activity and thickness of transversus abdominis (TrA), rectus abdominis (RA), lumbar multifidus (LM) and quadriceps muscles will be evaluated to evaluate muscle function. Muscle activity will be evaluated using surface electromyography (EMG) (Neuro-MEP, Ivanovo, Russia) and muscle thickness will be evaluated using ultrasound (LOGIQ P9, GE Healthcare, USA).
COPD Assessment Questionnaire | September 2024, July 2026
  The COPD Assessment Test (CAT) will be used to assess health status impairment in individuals with COPD. The CAT is an eight-item test consisting of questions that evaluate the severity of symptoms such as dyspnea, cough, and sputum production and the impact of the disease on daily life. It is recommended that the minimal clinical significance is a change of 2 points.
Timed up and go test | September 2024, July 2026
  The Timed Up and Go Test (TUG) will be used for the balance assessment of individuals participating in the study. TUG is a frequently used, easily applicable, valid and reliable, performance-based functional mobility and balance test that evaluates dynamic balance in the clinic. It has been shown that dynamic balance impairment in COPD is associated with inadequate oxygenation and peripheral muscle weakness. Individuals who complete the test in 12 seconds or more have a risk of falling
Functional reach test | September 2024, July 2026
  Functional reach test will be used for the balance assessment of individuals participating in the study. Individuals who can reach 25 cm and more have a low risk of falling. Individuals who can reach between 15-25 cm have a 2 times higher risk of falling than normal. Individuals who can reach 15 cm and below have a 4 times higher risk of falling than normal. Individuals who cannot reach at all have an 8 times higher risk of falling than normal.
St George Health Questionnaire | September 2024, July 2026
  St. George's Respiratory Questionnaire (SGRQ), a seventy-six-item health-related quality of life assessment questionnaire, will be used to assess the quality of life of the subjects.The result values are between 0 and 100 and the higher the value, the greater the degree to which the patient's quality of life is affected by the disease.
Hospital Anxiety and Depression Scale | September 2024, July 2026
  The Hospital Anxiety and Depression (HAD) scale will be used to determine the anxiety and depression levels of individuals participating in the study. This scale is a self-report scale that includes anxiety and depression subscales and consists of 14 items, seven of which investigate depression and seven of which investigate anxiety levels.The cut-off point for the anxiety subscale of the HAD Turkish form was found to be 10 and the cut-off point for the depression subscale was found to be 7. Patients who score above these points can be considered as a risk group. Anxiety and depression score 07: normal, 8-11: borderline, >11: anxiety and depression.
Six Minute Walk Test (6MWT) | September 2024- July 2026
  6MWT will be used to evaluate the exercise capacities of individuals who will participate in the study. The individuals' walking distance and cardiac parameters during the test will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)